CLINICAL TRIAL: NCT00064597
Title: National Institute of Child Health and Human Development Fetal Cell Isolation Study (NIFTY)
Brief Title: Noninvasive Prenatal Diagnosis: Using Fetal Cells From Maternal Blood
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: NICHD-NIFTY; 1N01HD43201; 1N01HD43202; 1N01HD43203; 1N01HD43204
Record Dates: First submitted 2003-07-10; First posted 2003-07-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Chromosome Disorders
Keywords: Fetal cells; Prenatal diagnosis; Cytogenetic disorders; Chromosomal disorders; Single gene mutation detection; Abnormal serum marker profile; Fluorescence activated cell sorting (FACS); Magnetic activated cell sorting (MACS); Fluorescence in situ hybridization (FISH); Chromosomal disorders of the fetus; Single gene defects of the fetus
MeSH Terms: conditions — Chromosome Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This purpose of this study is to develop noninvasive methods of prenatal diagnosis. Fetal cells can be found in maternal blood. This study is designed to isolate these fetal cells from a sample of the pregnant woman's blood and use those cells to test for fetal chromosome abnormalities.

DETAILED DESCRIPTION:
Fetal cells can be recovered from maternal blood, suggesting that noninvasive prenatal diagnosis is possible. However, recovery and analysis of fetal cells from maternal blood is complex and sensitivity is low because of the rarity of these cells in the maternal circulation. This study was designed to develop a noninvasive, safe, relatively inexpensive, and accurate technique for the prenatal diagnosis of genetic disorders in the first trimester.

The study included a systematic evaluation of variables involved in separating and enriching fetal cells isolated from maternal blood through fluorescence activated cell sorting (FACS) and magnetic activated cell sorting (MACS) followed by fluorescent in situ hybridization (FISH) with chromosome-specific DNA probes. The results of these tests were compared to those obtained from amniocentesis or chorionic villus sampling (CVS) on the same women. No clinical decision was made based on the results of the experimental diagnostic/screening technique.

Even if the biological risks associated with reproductive genetic technologies are reduced, it is possible that other risks (or benefits) are associated with the procedures. Some of these factors may be: increased or diminished maternal anxiety, increased adjustment or maladaption to the pregnancy, increased feelings of coercion to undertake the procedure, and increased or decreased comfort with reproductive decision-making. The study also assessed whether there were any nonbiological or psychological effects on the women undergoing prenatal diagnostic testing.

After the first five years of the study, preliminary analysis of the data showed that the sensitivity of aneuploidy detection using fetal cell analysis from maternal blood is comparable to single marker prenatal serum screening, but technological advances are needed before fetal cell analysis has clinical application as part of a multiple maker method for noninvasive prenatal screening. Target cell recovery and fetal cell detection were better using MACS than with FACS. The detection rate of finding at least one aneuploid cell in cases of fetal aneuploidy was 74.4%.

ELIGIBILITY:
Inclusion Criteria

* Pregnant
* Abnormal serum marker profile (alpha-fetoprotein, hCG, estriol)
* Ultrasound abnormalities of the fetus
* Any high risk indicator for aneuploidy as determined by physician

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3500
Dates: Start 1987-12; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Laird Jackson, MD, Principal Investigator; Diana Bianchi, MD, Principal Investigator; Mark Evans, MD, Principal Investigator; Sherman Elias, MD, Principal Investigator
Locations (5):
- United States (5):
  - University of Illinois at Chicago, Chicago, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Bischoff FZ, Hahn S, Johnson KL, Simpson JL, Bianchi DW, Lewis DE, Weber WD, Klinger K, Elias S, Jackson LG, Evans MI, Holzgreve W, de la Cruz F. Intact fetal cells in maternal plasma: are they really there? Lancet. 2003 Jan 11;361(9352):139-40. doi: 10.1016/S0140-6736(03)12191-5. PMID 12531583
- [Background] Bianchi DW, Simpson JL, Jackson LG, Elias S, Holzgreve W, Evans MI, Dukes KA, Sullivan LM, Klinger KW, Bischoff FZ, Hahn S, Johnson KL, Lewis D, Wapner RJ, de la Cruz F. Fetal gender and aneuploidy detection using fetal cells in maternal blood: analysis of NIFTY I data. National Institute of Child Health and Development Fetal Cell Isolation Study. Prenat Diagn. 2002 Jul;22(7):609-15. doi: 10.1002/pd.347. PMID 12124698
- [Background] Bianchi DW. Prenatal exclusion of recessively inherited disorders: should maternal plasma analysis precede invasive techniques? Clin Chem. 2002 May;48(5):689-90. No abstract available. PMID 11978594
- [Background] Bohmer RM, Stroh HP, Johnson KL, LeShane ES, Bianchi DW. Fetal cell isolation from maternal blood cultures by flow cytometric hemoglobin profiles. Results of a preliminary clinical trial. Fetal Diagn Ther. 2002 Mar-Apr;17(2):83-9. doi: 10.1159/000048014. PMID 11844911
- [Background] Lee T, LeShane ES, Messerlian GM, Canick JA, Farina A, Heber WW, Bianchi DW. Down syndrome and cell-free fetal DNA in archived maternal serum. Am J Obstet Gynecol. 2002 Nov;187(5):1217-21. doi: 10.1067/mob.2002.127462. PMID 12439507